CLINICAL TRIAL: NCT04902755
Title: French Version of the Short Form of Neurogenic Bladder Symptom Score: Cross-Cultural Adapta-tion and Validation.
Brief Title: French Version of the Short Form of Neurogenic Bladder Symptom Score
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Clinical Professor, Pierre and Marie Curie University
Other Study IDs: GREEN NBSS SF
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Neurogenic Bladder
Keywords: Questionnaire; Neurogenic bladder; multidimensionnal; LUTS
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — validation of the French linguistic version and the cross-cultural adaptation of the NBSS-SF.

SUMMARY:
Lower urinary tract symptoms (LUTS) are frequent in worldwide population. In neurogenic condition, LUTS can occur from beginning of neurologic disease (SCI, MS) or during its progression (MS). Neurogenic bladder may be responsible for upper urinary tract complications such as urinary tract infection or renal failure. It can also decrease quality of life and have an important socio-economic impact. For the last few years, patient-reported outcomes (PRO) have been the main way to assess functional urinary symptoms such as urinary incontinence or overactive bladder. Fortunately, Welk and al. developed and validated a new questionnaire in 2013 to allow a multimodal evaluation of LUTS specifically designed for a neurogenic population. The Neurogenic Bladder Symptom Score (NBSS) is composed of 24 items and explores 3 domains (urinary incontinence, bladder storage and voiding, consequences). In addition, NBSS includes two additional questions related to bladder management and quality of life. In 2020, Welk and al. developed a short version of NBSS (NBSS-SF), composed of 10 items exploring the 3 same domains as the NBSS original long version. However, there is no French-validated multi-dimensional questionnaire specifically assessing neurogenic LUTS, the USP questionnaire being a generic tool (Urinary Symptoms Profile (USP)).

The objective of our study was to validate the French linguistic version and the cross-cultural adaptation of the NBSS-SF.

METHODS:

The investigators conducted a prospective monocentric study between June and October 2020 in our neuro-urology clinic.

Step 1, translation and back-translation:

With the author's agreement, two bilingual translators (fluent in English and native French) created a French version of the NBSS. Both versions were combined and disagreement in wording or item redaction were resolved to maintain a better understanding. Next step was the back-translation with an native English translator.

Then, a bilingual expert committee, composed by urologists and neuro-urologists, compared the different versions to create a pre-final version of the questionnaire. Cross-cultural equivalence with analysis of the semantic, idiomatic, conceptual, and empirical equivalence of the source and pre-final versions of the NBSS-Short Form have been validated by the expert committee.

Step 2, Pilot study : n = 30 subjects. During this pilot study, acceptability and understanding were evaluated. Participant had to answer with a 3 level Likert scale (A: perfectly; B: good; C: poor) for each item. Comprehension and acceptation were considered as good if they answered A or B. All difficulties and remarks were collected to incorporate these comments in the final version after validation by a panel of experts.

Step 3, Validation stud:

To perform validation study, the investigators used the same inclusion criteria than Welk and al. and included patients with a neurogenic bladder due to multiple sclerosis (MS), spinal cord injury (SCI) or other neurologic condition such as spina bifida or Parkinson disease.

Validation study was performed to determine the psychometric properties of the questionnaire.

The investigators calculated the Cronbach's α coefficient, a measure of internal consistency (reliability) ranging from 0-1, with a coefficient greater than 0.7 considered as very good. The NBSS-short form is composed of 2 first items (covering quality of life and bladder management) and 8 items covering 3 subdomains (items 3, 4, 5 for urinary incontinence, items 6, 7, 8 for storage and voiding) and finally 2 items covering the consequences. The investigators calculated a Cronbach's α coefficient for each subscale and a coefficient for the whole questionnaire.

For test-retest reliability, the intraclass correlation coefficient (ICC) has been used. An ICC greater than 0.7 is considered as a good test-retest reproducibility. Participants completed the final version of the questionnaire and they had to mail the second questionnaire within 7 to 14 days. As this second questionnaire was completed at home, all participants were called to avoid missing data.

Correlations were computed between NBSS-SF scores obtained overall and for each domain on two different occasions, separated by a 7-14-day interval.

ELIGIBILITY:
Inclusion Criteria:

* patients with a neurogenic bladder
* Understand and read French language

Exclusion Criteria:

* recent urological surgery
* recent urinary tract infection
* treatment modification during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total, 105 patients were included with 59 women (56%) and mean age was 53 years. They were affected by a variety of neurological disorders: 58 (55%) had Multiple Sclerosis, 17 (16%) had a Spinal Cord Injury, and 30 (29%) had other neurological conditions such as Parkinson's disease, spina bifida or cauda equina syndrome
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
French translation of NBSS SF | 14 days
  good or very good psychometric properties of the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Neurourology department, Hopital tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided